CLINICAL TRIAL: NCT03779217
Title: BREast Density in Premenopausal Women is Predictive of CARdiovascular Outcomes at 10 Years of Follow-up: the BRECARD Study
Brief Title: Breast Disease and Cardiovascular Disease
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Celestino Sardu, medical doctor, University of Campania Luigi Vanvitelli
Other Study IDs: SecondUNI 17.12.2018
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Cardiovascular Diseases; Ischemic Heart Disease
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Ischemia | interventions — Mammaplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- group A: In this group there are women in that the mammography shows a breast represented by 80% of adipose tissue and less than 20% by fibro-glandular tissue.
  Interventions: Other: screening mammography; Procedure: mastoplasty and breast fat excission
- group B: In this group there are women in that the mammography shows a breast represented by adipose tissue in the range of 50-75% and for the rest by fibro-glandular tissue
  Interventions: Other: screening mammography; Procedure: mastoplasty and breast fat excission
- group C: In this group there are women in that the mammography shows a breast represented by adipose tissue in the range 25-50% and the rest is from fibro-glandular tissue.
  Interventions: Other: screening mammography; Procedure: mastoplasty and breast fat excission
- group D: In this group there are women in that the mammography shows a breast represented by almost entirely fibro-ghiandular tissue.
  Interventions: Other: screening mammography; Procedure: mastoplasty and breast fat excission

INTERVENTIONS:
Other: screening mammography — As indicated by international guidelines authors will perform screening mammography in all asymptomatic women.
Procedure: mastoplasty and breast fat excission — As indicated by guidelines, and in accordance to the breast surgery reduction criteria, the authors will practice a surgical intervention of mastoplasty. During the mastoplasty, authors will remove the breast fat tissue.

SUMMARY:
Cardiovascular disease (CVD) occurs less frequently in women than in juvenile men.Frequently the estrogen deficiency associated with the menopausal state affects cardiovascular outcomes. In fact, in the post-menopausal state, even younger women may experience an increase in the rate of ischemic heart disease (IHD). On the other hand, CVD may also occur in premenopausal young women, due to not well known and/or not clearly investigated mechanisms. In addition, pre-menopausal women with IHD show atypical symptoms and more frequently myocardial infarction vs. angina pectoris. In detail, in these patients IHD is frequently due to mono-vessel coronary heart disease, and to the presence of cardiovascular risk factors such as hypertension, hyperlipidemia and type 2 diabetes. So, it is clear that all these pro-atherogenic risk factors which lead to IHD in women, are significantly lower in the pre-menopausal vs. post-menopausal patients. However, the causes leading to IHD and acute coronary events in pre-menopausal women remain poorly understood and poorly investigated, and these factors might be different from the traditional coronary risk factors evident in the general population. In this context, recently some authors have shown that subcutaneous abdominal fat affects cardiovascular performance at 1 year of follow-up in patients with normoglycemia vs. pre-diabetic. Therefore, here authors can hypothesize that in a population of female subjects, the fat tissue present in the mammary gland and the different degrees of mammary adipocyte infiltration can somehow invalidate the number of cardiovascular events in women of childbearing age. In detail, the different distribution of adipose tissue in the mammary gland can influence the density of the breast, as studied by mammographic examination, which is used to divide breast density into 4 different categories:

* Category A: the breast is represented by 80% of adipose tissue and less than 20% by fibro-glandular tissue.
* Category B: the breast is represented by adipose tissue in the range of 50-75% and for the rest by fibro-glandular tissue.
* Category C: the breast is represented by fatty tissuein the range 25-50% and the rest is from fibro-glandular tissue
* Category D: the breast is represented by almost entirely fibro-glandular tissue.

Therefore, in the present study authors correlated the 4 different breast categories with CVD and 10-year follow-up IHD in women of child-bearing age. In fact, according to authors' opinion, a breast with higher fat density (category A) might influence the number of adverse cardiovascular events at 10-year follow-up in asymptomatic women. Thus, pre-menopausal women with breast tissue in category A ("fatty breast") as compared to women with prevalence of fibro-glandular tissue ("non-fatty breast") may have a higher frequency of adverse cardiac ischemic events at 10 years of follow-up.

On the other hand, the molecular pathways implied in worse CVD in these cohorts of women are not fully investigated.

Furthermore, the authors aimed to investigate the expression of inflammatory cytokines and sodium glucose transporter 2 (SGLT2) protein expression, as markers of over-inflammation, at level of breast gland in these cohorts of women. Thus, these markers were analyzed in the breast fat tissue excissed from the fatty vs. non-fatty breast women.

ELIGIBILITY:
Inclusion Criteria:

* patients with indication to receive a screening MiD, patients without breast cancer diagnosis (previous or recent diagnosis), pre-menopausal status, without inflammatory chronic disease and other neoplastic diseases. Patients without previous history of cardiovascular and cerebrovascular adverse events. Patients with indication to receive a breast reduction surgery (relief of physical pain and discomfort associated with heavy, pendulous breasts; complain of chronic back and neck pain, headaches, shoulder pain, deep bra-strap grooves, and rashes beneath both breasts; breast chronically painful as well, evidence of upper extremity neuropathy and postural changes, along with intertrigo, maceration, irritation, rashes, and other dermatologic manifestations; difficulty with many forms of exercise and the inability to find properly fitting clothe; patients that received a full package of supportive care, advising on weight loss and managing pain, physiotherapy and assessment for thoracic / shoulder girdle discomfort).

Exclusion Criteria:

* aged < 18 years, patients without indication to receive a screening MiD, patients with breast cancer diagnosis (previous or recent diagnosis), menopausal status, inflammatory chronic disease, other neoplastic diseases; previous history of cardiovascular and cerebrovascular adverse events.

Ages: 18 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: The study population will include asymptomatic women without neoplastic breast disease and other neoplastic diseases. These patients at enrollment did not have previous history of cardiovascular and cerebrovascular adverse events. At enrollment all women did not have a diagnosis of menopausal status.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2008-01-02 (Actual); Primary Completion 2021-01-02 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
myocardial infarction | 10 years
  Authors will evaluated for all follow up duration the number of myocardial infarction

CONTACTS AND LOCATIONS:
Locations (1):
- Raffaele Marfella, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sardu C, Gatta G, Pieretti G, Viola L, Sacra C, Di Grezia G, Musto L, Minelli S, La Forgia D, Capodieci M, Galiano A, Vestito A, De Lisio A, Pafundi PC, Sasso FC, Cappabianca S, Nicoletti G, Paolisso G, Marfella R. Pre-Menopausal Breast Fat Density Might Predict MACE During 10 Years of Follow-Up: The BRECARD Study. JACC Cardiovasc Imaging. 2021 Feb;14(2):426-438. doi: 10.1016/j.jcmg.2020.08.028. Epub 2020 Oct 28. PMID 33129736